CLINICAL TRIAL: NCT04145024
Title: Giessen Pulmonary Hypertension Registry and Biobank
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: 2001
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Pulmonary arterial hypertension: Group 1 PH
- Pulmonary hypertension due to left heart disease: Group 2 PH
- Pulmonary hypertension due to lung disease: Group 3 PH
- Chronic thromboembolic pulmonary hypertension: Group 4 PH
- Miscellaneous: Group 5 PH
- Exclusion PH: Patient with invasively excluded PH

SUMMARY:
Giessen Pulmonary Hypertension Registry and Biobank

DETAILED DESCRIPTION:
Long-term transplant-free survival and its determinants will be investigated in patients with Pulmonary Hypertension (diagnosed by right heart catheterization) within a prospective registry at a single referral center in Giessen, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Right heart catheterization for PH diagnosis in Giessen

Exclusion Criteria:

* informed consent missing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes patients referred to our tertial PH expert center in Giessen with suspected PH.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1993-07 (Actual); Primary Completion 2035-07-15 (Estimated); Study Completion 2036-01-15 (Estimated)

PRIMARY OUTCOMES:
Survival | Up to 20 years after enrollment
  Transplant-free survival of PH patients

CONTACTS AND LOCATIONS:
Overall Officials: Khodr Tello, MD, Principal Investigator — University Clinics of Giessen and Marburg
Locations (1):
- Department of Intermal Medicine - Universities of Giessen and Marburg Lung Center, Giessen, Germany

REFERENCES:
- [Result] Gall H, Felix JF, Schneck FK, Milger K, Sommer N, Voswinckel R, Franco OH, Hofman A, Schermuly RT, Weissmann N, Grimminger F, Seeger W, Ghofrani HA. The Giessen Pulmonary Hypertension Registry: Survival in pulmonary hypertension subgroups. J Heart Lung Transplant. 2017 Sep;36(9):957-967. doi: 10.1016/j.healun.2017.02.016. Epub 2017 Feb 17. PMID 28302503